CLINICAL TRIAL: NCT00327756
Title: An Investigation Examining the Evidence for Mitochondrial Dysfunction in the Pathophysiology and Treatment of Bipolar Disorder
Brief Title: Mitochondrial Dysfunction in the Pathophysiology and Treatment of Bipolar Disorder
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Carlos A. Zarate, M.D./National Institute of Mental Health, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 060162; 06-M-0162
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2009-05

CONDITIONS: Bipolar Affective Disorder; Depression
Keywords: Depression; Magnetic Resonance Spectroscopy; Mitochondrial Enhancer; Manic Depressive; Bioenergetics; Bipolar Disorder; Manic Depression
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Coenzyme Q10

SUMMARY:
This study will examine whether mitochondrial function is impaired in patients with bipolar disorder. Mitrochondria are small organelles inside the cell that are responsible for energy production. Recent studies in animals and humans suggest that abnormalities of mitrochondria may be involved in bipolar depression. The study will also examine whether the food supplement Coenzyme Q10 (CoQ10) improves mitochondrial function and symptoms such as depressed mood, low energy, anxiety or slowness in thinking and movements in bipolar patients. CoQ10 has been used to increase cell energy production and as an antioxidant. It has had some benefit in patients with Parkinson's disease and migraine and in prolonging survival in patients with cancer and heart failure.

Patients 18-65 years of age with bipolar disorder who are currently in a depressive episode of at least 4 weeks duration may be eligible for this study. The study has four phases, as follows:

Phase I: Medication Withdrawal

Patients taper off all psychotropic medications, usually over 1 to 2 weeks.

Phase II: Baseline Evaluation

After being off all medication for about 2 weeks, patients undergo the following procedures:

* Magnetic resonance imaging (MRI) and magnetic resonance spectroscopy (MRS). The two procedures are performed in an MRI scanner. Both tests use a strong magnetic field and radio waves to obtain images that provide information on brain anatomy and chemistry.
* Blood tests to assess mitochondrial function isolated from blood cells.
* Skin biopsy for tests of mitochondria. A small sample of skin tissue 5 x 5 millimeters is surgically removed.

Phase III: Administration of CoQ10 or Placebo

Participants are randomly assigned to take either CoQ10 or placebo (an inactive look-alike substance) twice a day by mouth. While taking the study medication, patients have the following procedures periodically:

* Rating scales for anxiety and depression and adverse events.
* Check of vital signs.
* Blood and urine sample collections.

Phase IV: Study Completion

At the end of the 8 weeks of treatment, patients have a physical examination and electrocardiogram, and the procedures in phase II are repeated. Participants may then receive short-term treatment (up to 12 weeks) with medications for bipolar depression, followed by referred to a community physician for long-term treatment.

...

DETAILED DESCRIPTION:
Bipolar affective disorder is a common, severe, chronic and often life-threatening illness. The depressive phase contributes to the majority of morbidity and mortality in this illness. Impairments in physical and social functioning resulting from depression are often as severe as other chronic medical illnesses. Few of the treatments in use have resulted from an understanding of the pathophysiology of bipolar disorder. Undoubtedly, a greater understanding of the pathophysiology of bipolar disorder will lead to improved treatments.

Current theories of depression suggest that mood disorders are associated with impairments of cellular resilience and structural plasticity possibly a result of abnormal cellular energy metabolism. Studies with Magnetic Resonance Spectroscopy (MRS) in bipolar subjects show reduced brain intracellular pH and reduced ATP. Cellular energy generated by mitochondrial oxidative phosphorylation from glucose via the electron transport chain is stored as ATP, which provide neurons and glia with energy required to maintain their function. Mitochondrial dysfunction and its inability to compensate for increase in ATP demand might lead to impaired cellular resilience believed to be involved in the pathophysiology of bipolar disorder. Abnormal regulation of nuclear genes coding for mitochondrial proteins in the hippocampus of bipolar subjects provides further evidence of mitochondrial dysfunction in bipolar disorder.

Coenzyme Q10 (CoQ10) is an essential cofactor in the mitochondrial electron transport chain necessary for cellular energy generation. Exogenous administration of CoQ10 attenuates ATP depletion and has anti-oxidant properties. In light of the above evidence, we hypothesize that bipolar disorder is associated with mitochondrial dysfunction as evidenced by impaired brain energy metabolism and that administration of CoQ10, a mitochondrial enhancer, will restore mitochondrial function. To accomplish these objectives, we will compare mitochondrial functions in bipolar depressed subjects to 26 healthy controls matched for age, gender and BMI. Measures of mitochondrial function will include brain lactate levels (a product of anaerobic glycolysis) with H+ MRS, 2) assays of mitochondrial function in cultured fibroblasts and platelets, and 3) gene expression of mitochondrial and nuclear genes using a cDNA Microarray. Further, subjects with bipolar depression, ages 18 to 65 will be randomized to either CoQ10 (300-1200 mg/day) or placebo in a double-blind placebo controlled trial for a period of 8 weeks. Measures of mitochondrial function will be compared between subjects randomized to placebo or CoQ10 at baseline and at the end of the 8-week trial.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Male or female subjects, 18 to 65 years of age.
* Female subjects of childbearing potential must be using a medically accepted means of contraception.
* Each subject must understand the nature of the study and must sign an informed consent document.
* Subjects must fulfill the criteria for Bipolar disorder depressed without psychotic features including rapid cycling as defined in DSM-IV based on clinical assessment and confirmed by structured diagnostic interview SCID-P.
* Subjects must have an initial score at Visit 1 and Visit 2 of at least 16 on the MADRS
* In bipolar II disorder, subjects must have experienced, in the opinion of the investigator, at least two previous hypomanic and two major depressive episodes as defined in DSM-IV.
* Current major depressive episode at least 4 weeks in duration.

EXCLUSION CRITERIA:

* Subjects who are currently on a mood stabilizer for maintenance treatment and are benefiting from it.
* Current diagnosis of primary anxiety disorder necessitating treatment (subjects with OCD will be excluded).
* Presence of psychotic features
* Participation in a clinical trial of another investigational drug within 1 month prior to study entry (Visit 1).
* Female subjects who are either pregnant or nursing.
* Serious, unstable illnesses including hepatic, renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease), endocrinology, neurological, immunologic, or hematological disease.
* Subjects diagnosed with a mitochondrial disorder.
* Subjects taking other putative mitochondrial enhancers (e.g., vitamin E, carnitine, creatine, Vit complex B, pramipexole; see Appendix B) by the time of randomization (Visit 2).
* Subjects taking Statins
* Subjects with Diabetes Mellitus (Type I and Type II)
* Subjects with a history of clotting disorders or needing anticoagulants e.g. warfarin.
* Subjects with history of deep vein thrombosis or the following risk factors for DVTs, smoking and/or contraceptives (30 days before Visit 2).
* Subjects with uncorrected hypothyroidism or hyperthyroidism.
* Subjects with one or more seizures.
* Documented history of hypersensitivity or intolerance to CoQ10.
* DSM-IV substance abuse (except caffeine) within the past 12 months, 1 month for nicotine.
* DSM-IV lifetime substance dependence (except caffeine).
* Treatment with an injectable depot neuroleptic within less than one dosing interval prior to Visit 2.
* Treatment with a reversible MAOI, guanethidine, or guanadrel within 1 week prior to Visit 2.
* Treatment with fluoxetine within 6 weeks prior to Visit 2.
* Treatment with any other concomitant medication 1 day prior to Visit 2.
* Treatment with clozapine or ECT within 1 month prior to Visit 2.
* Judged clinically to be at serious suicidal risk.

Healthy Control Sample: Twenty-six subjects (ages 18-65) who do not meet criteria for any major medical or psychiatric disorder (using SCID -NP) will undergo imaging and mitochondrial assay part of the study and serve as control group. Control subjects will be matched to bipolar subjects for age, gender, Body Mass Index (BMI) plus or minus 2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-05; Primary Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Compare brain lactate levels between healthy controls and subjects with bipolar depression and assess in subjects w/bipolar depression the effect of of CoQ10 admin compared to placebo on the brain lactate signal obtained w/MRS w/photic stimulation. | 8 weeks

SECONDARY OUTCOMES:
To determine the antidepressant efficacy of CoQ10 compared to placebo in depressed subjects w/bipolar disorder by using the mean change in MADRS total score pre- and post-study. | 8-weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Arias-Mendoza F. In vivo magnetic resonance spectroscopy in the evaluation of mitochondrial disorders. Mitochondrion. 2004 Sep;4(5-6):491-501. doi: 10.1016/j.mito.2004.07.034. Epub 2004 Sep 30. PMID 16120408
- [Background] Baker SK, Tarnopolsky MA. Targeting cellular energy production in neurological disorders. Expert Opin Investig Drugs. 2003 Oct;12(10):1655-79. doi: 10.1517/13543784.12.10.1655. PMID 14519086
- [Background] Bertolino A, Frye M, Callicott JH, Mattay VS, Rakow R, Shelton-Repella J, Post R, Weinberger DR. Neuronal pathology in the hippocampal area of patients with bipolar disorder: a study with proton magnetic resonance spectroscopic imaging. Biol Psychiatry. 2003 May 15;53(10):906-13. doi: 10.1016/s0006-3223(02)01911-x. PMID 12742678